CLINICAL TRIAL: NCT02583139
Title: The Effect and Meaning of Designed Music Narratives on Anticipatory, Acute, and Delayed Side Effect of Chemotherapy in Children (7-12 Years) With Cancer: a Randomized Controlled Multisite Study
Brief Title: Designed Music Narratives for the Reduction of Side Effects of Chemotherapy in Children (7-12 Years) With Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Danish Cancer Society (Other); Børnecancerfonden (Other); Ronald McDonalds Børnefond (Other); TrygFonden, Denmark (Industry)
Responsible Party: Principal Investigator, Ilan Sanfi, Music therapist, PhD, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MF-Cancer-Children-1
Record Dates: First submitted 2015-02-03; First posted 2015-10-22 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Cancer; Chemotherapy-induced Nausea and Vomiting; Effects of Chemotherapy
Keywords: Children, Moderate and/or highly emetogenic chemotherapy
MeSH Terms: conditions — Neoplasms; Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music Narrative Group (Experimental): Prescribed medical/chemotherapy treatment plus standard care + Designed Music Narratives
  Interventions: Behavioral: Designed Music Narratives
- Control Group (No Intervention): Prescribed medical/chemotherapy treatment plus standard care

INTERVENTIONS:
Behavioral: Designed Music Narratives — Four music narratives for children each comprising an introductory relaxation exercise, a resource-oriented narrative including guided imagery suggestions and relaxing nature scenarios plus especially composed music.
  The narrative and music reflect and support each other.
  Arms: Music Narrative Group

SUMMARY:
The purpose of this study is to determine whether a specially-designed music-narratives are effective in reducing side effects of chemotherapy in 7- to 12-year-olds with cancer.

DETAILED DESCRIPTION:
(Will be added later)

ELIGIBILITY:
1. Children at the ages 7-12
2. Four or five (dependent on their overall plan of medical treatment) consecutive courses of chemotherapy administrated at the involved child cancer units and (administered) over a period of minimum 24 hours incl. hydration with assumed moderate to severe nausea and vomiting.

   The specific type of chemotherapy may vary across the four/five consecutive courses but shall include one of the following moderate and/or highly emetogenic types of chemotherapy:

   Moderate emetogenic chemotherapy:
   * Carboplatin
   * Cyclophosphamide <1500 mg/m2
   * Cytarabine >1 g/m2
   * Daunorubicin
   * Doxorubicin
   * Epirubicin
   * Idarubicin
   * Ifosfamide
   * Mitoxantrone
   * Methotrexate >1000 mg/m2

   Highly emetogenic chemotherapy:
   * Cisplatin >25 mg/m2
   * Cyclophosphamide >1500 mg/m2
   * Dacarbazine
3. Understand Norwegian/Danish
4. Parents must be able to read and understand Norwegian/Danish

   * No significant hearing impairment
   * Written and verbal informed consent from both possessors of the custody
   * Verbal informed consent from child/participant

Exclusion Criteria:

* Previous and/or acute psychiatric diagnosis
* Cognitive and mental deficits or impaired functioning

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2014-08; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Duration (minutes) of Acute Nausea | Registered the two first evenings within the first 32 hours after onset of chemotherapy during 5th cycle of chemotherapy after enrolment in study
  Self-reported duration og nausea in minutes within the first 32 hours after onset of chemothera

SECONDARY OUTCOMES:
Intensity of Acute Nausea as measured by the Visual Analogue Scale | Registered the two first evenings within the first 32 hours after onset of chemotherapy during 5th cycle of chemotherapy after enrolment in study
  Self-reported intensity of nausea, calculated as the average of the two measurements
Distress regarding Acute Nausea as measured by the Visual Analogue Scale | Registered the two first evenings within the first 32 hours after onset of chemotherapy during 5th cycle of chemotherapy after enrolment in study
  Self-reported distress regarding nausea, calculated as the average of the two measurements
Amount (mg/m2) of Nausea Reducing Medicine Consumed | During admission (an expected average of 3 days) and the first three days after discharge regarding 5th cycle of chemotherapy after enrolment in study
Multiple Acute Side Effects of Chemotherapy as measured by the Memorial Symptom Assessment Scale | Registered the two first evenings within the first 32 hours after onset of chemotherapy during 5th cycle of chemotherapy after enrolment in study
  Self-reported side effects, calculated as the average of the two measurements. The Memorial Symptom Assessment Scale is a self-report composite measure that measures bodily and psychological symptoms of side effects
Numbers of Acute Vomiting | Registered the two first evenings within the first 32 hours after onset of chemotherapy during 5th cycle of chemotherapy after enrolment in study
  Self-reported numbers of vomiting during the first 32 hours
Duration (minutes) of Acute Pain | Registered the two first evenings within the first 32 hours after onset of chemotherapy during 5th cycle of chemotherapy after enrolment in study
  Self-reported duration of acute pain in minutes within the first 32 hours after onset of chemotherapy
Acute Pain Intensity as measured by the Visual Analogue Scale | Registered the two first evenings within the first 32 hours after onset of chemotherapy during 5th cycle of chemotherapy after enrolment in study
  Self-reported intensity of pain, calculated as the average of the two measurements
Number of Days to Absolute Neutrophil Count Recovery (ANCR) defined as ANCR ≥ 0.5 x 109/L | Time to Event: Measured Day 1 in 5th cycle of chemotherapy after enrolment in study - until first day with ANC ≥ 0.5 x 109/L after the nadir period (an expected average of 9-15 days)
  Number of days before the immune system recovers after chemotherapy. In the study, Absolute Neutrophil Count Recovery (ANCR) is defined as ANCR ≥ 0.5 x 109/L. In addition, if no nadir < 0.5 x 109/L occurs the period is 0 (zero)
Duration (minutes) of Acute Fatigue | Registered the two first evenings within the first 32 hours after onset of chemotherapy during 5th cycle of chemotherapy after enrolment in study
  Self-reported duration of acute fatigue in minutes within the first 32 hours after onset of chemotherapy
Distress of Acute Fatigue as measured by a 5-point Likert-type Scale | Registered the two first evenings within the first 32 hours after onset of chemotherapy during 5th cycle of chemotherapy after enrolment in study
  Self-reported Distress regarding Acute Fatigue, calculated as the average of the two measurements
Appraised Food Intake and Appetite as measured by a 5-point Likert-type Scale | Registered the two first evenings within the first 32 hours after onset of chemotherapy during 5th cycle of chemotherapy after enrolment in study
  Self-reported appraised food intake, calculated as the average of the two measurements
Weight (kg) | Change between weight from during course 1 and course 5 after inclusion in study
Satisfaction with Applied Music Intervention as measured by a Likert-type Scale (participants in music group only) | Last day (i.e. expected 3rd or 4th day) of 5th cycle of chemotherapy after enrolment in study
  Self-report, registered once during 5th cycle of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Sanfi, PhD, Principal Investigator — Aarhus University Hospistal
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark